CLINICAL TRIAL: NCT06636747
Title: A Comparative Study of High Resolution DWI and Conventional DWI in Prostate
Brief Title: High Resolution Diffusion Weighted Imaging in Prostate
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-586
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Prostate Disease
Keywords: diffusion weighted imaging; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
hrDWI might be an alternative to cDWI for the prostate imaging.

1. increase the signal-to-noise ratio and contrast-to-noise ratio, yielding high-fidelity images with less noise in general
2. improve the diagnostic accuracy of PCa in particular than conventional DWI

DETAILED DESCRIPTION:
Magnetic Resonance Imaging (MRI) with the Prostate Imaging Reporting and Data System (PI-RADS) is a state-of-the-art strategy, not only for standardizing prostate MRI scanning, but also for PCa detection, diagnosis and staging. In PI-RADS score evaluation, diffusion weighted imaging (DWI) is an important component of the prostate MRI examination, which is considered to be the dominant sequence for the assessment of lesions in the peripheral zone (PZ) and is also regarded as the auxiliary sequence for the upgrade of lesions in the transitional zone (TZ). DWI reflects the random motion of water molecules, that should include high b-value images (at least b≥1400s/mm²) and an calculated ADC map. As the b-value increases, DWI enables detection of small changes because of better contrast between malignant and background tissue. Meanwhile, the problems arise. DWI is often plagued by poor spatial resolution, distortion, and artifacts, as well as decreased signal-to-noise ratio (SNR) and contrast-to-noise ratio (CNR). This is a major obstacle to the application, interpretation, and ultimate impact of prostate MRI. Improving the quality of DWI images would be helpful in lesion orientation and detection of small cancers.Recently, a novel denoising technique, that operating on repetitively acquired MRI data and only removing components that cannot be distinguished from zero-mean Gaussian distributed noise, has been proposed for acquisition of ultra-high resolution images. Recent studies have shown that ultra-high resolution images significantly improvements in temporal-SNR, the detection and reproducibility of stimulus-induced signal changes, and the accuracy of images. Based on reconstruction algorithms with trainable components, high resolution DWI (hrDWI) can increase the SNR and CNR, yielding high-fidelity images with less noise in general, and thus to improve the diagnostic accuracy of PCa in particular than conventional DWI (cDWI).Therefore, we made the hypothesis that hrDWI might be an alternative to cDWI for the prostate imaging. The purpose of this study includes two aspects: 1) compare objective and subjective image quality and lesion conspicuity of hrDWI with cDWI in prostate MRI; 2) test the non-inferiority of hrDWI in terms of PCa diagnosis against cDWI in a cohort of suspcious patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent standard MR scanning including T2WI, cDWI , hrDWI and respective calculated apparent diffusion coefficient (ADC) maps;
2. Complete clinical information.

Exclusion Criteria:

Men were excluded if they were using 5-alpha-reductase inhibitors at time of examination or has used such during the previous six months; or if they had a previous history of prostatic biopsy, prostatic surgery, or treatment for PCa

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men larger than 55 years old were eligible to participate if they had a clinical suspicion of PCa with no previous biopsy. This included those with elevated PSA (> 4 ng/ml), or with suspicious digital rectal examination findings, or with suspicious findings on ultrasound examination, or with a family history of PCa.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
image quality evaluation | 2024.01-2025.12
  objective and subjective image quality and lesion conspicuity

SECONDARY OUTCOMES:
prostate cancer diagnosis | 2024.01-2025.12
  the diagnostic accuracy of prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Fei-Yun Wu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Yu-Dong Zhang, Nanjing